CLINICAL TRIAL: NCT05197049
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Guselkumab Subcutaneous Induction Therapy in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Guselkumab Subcutaneous Therapy in Participants With Moderately to Severely Active Crohn's Disease
Acronym: GRAVITI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109125; CNTO1959CRD3004 (Other: Janssen Research & Development, LLC); 2020-006165-11 (EudraCT Number); 2023-504737-41-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab (Experimental): Participants will receive guselkumab (Dose 1) injection subcutaneously followed by guselkumab (Dose 2) injection subcutaneously.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab (Dose 1) injection subcutaneously followed by guselkumab (Dose 3) injection subcutaneously.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 3
- Group 3: Placebo (Placebo Comparator): Participants will receive placebo injection subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Guselkumab (Dose 1) will be administered by subcutaneous (SC) injection.
  Arms: Group 1: Guselkumab; Group 2: Guselkumab
Drug: Guselkumab Dose 2 — Guselkumab (Dose 2) will be administered by SC injection.
  Arms: Group 1: Guselkumab
Drug: Guselkumab Dose 3 — Guselkumab (Dose 3) will be administered by SC injection.
  Arms: Group 2: Guselkumab
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Group 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of guselkumab in participants with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease (CD) of at least 3 months in duration
* Have moderate to severe CD as assessed by CDAI, stool frequency, and abdominal pain score, and Simple Endoscopic Score for Crohn's disease (SES-CD).
* Demonstrated intolerance or inadequate response to conventional or to biologic therapy for CD

Exclusion Criteria:

* Current diagnosis of ulcerative colitis or indeterminate colitis
* Complications of Crohn's disease that require surgical intervention or confound efficacy assessments
* Unstable doses of concomitant Crohn's disease therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2028-10-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (342):
- United States (76):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Advanced Gastro P.C, Chandler, Arizona
  - Reliance Research, Scottsdale, Arizona
  - Moore Clinical Trials, LLC, Little Rock, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Om Research LLC, Lancaster, California
  - United Gastroenterologists, Los Alamitos, California
  - Paul Wallace MD, Los Angeles, California
  - Clinnova Research, Orange, California
  - Digestive System Healthcare, Pasadena, California
  - Northshore Gastroenterology Research, LLC, San Diego, California
  - Clinical Applications Laboratories, Inc, San Diego, California
  - Santa Maria Gastroenterology, Santa Maria, California
  - Clinical Research of California, Walnut Creek, California
  - Amel Med LLC Research, Grand Junction, Colorado
  - Western Connecticut Health Network/Danbury Hospital, Danbury, Connecticut
  - Gastroenterology Associates of SW Florida, Clearwater, Florida
  - Pioneer Research Solutions Inc., Coconut Creek, Florida
  - Omega Research Consultants, DeBary, Florida
  - Harmony Medical Research Institute, Inc., Hialeah, Florida
  - Central Florida Gastro Research, Kissimmee, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Center for Digestive Health, Orlando, Florida
  - Central Florida Internists, Orlando, Florida
  - Synergy Clinical Research, St. Petersburg, Florida
  - Atlanta Gastroenterology Specialists, PC, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Atlanta Center For Gastroenterology, Decatur, Georgia
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - Gastroenterology Consultants, Roswell, Georgia
  - USF Asthma, Allergy, Immunology Clinical Research Unit, Boise, Idaho
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Lemah Creek Clinical Research, Oakbrook Terrace, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - BVL Clinical Research, Leawood, Kansas
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Institute for Digestive Health and Liver Disease, Baltimore, Maryland
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Digestive Health Specialists PC, Chelmsford, Massachusetts
  - FC Research, LLC, South Dartmouth, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Detroit Clinical Research Center, Livonia, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Smart Medical Research, Jackson Heights, New York
  - Crystal Run Healthcare LLP, Middletown, New York
  - New York Gastroenterology Associates, New York, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - A1 Clinical Network, Queens, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Gastroenterology Associates of the Piedmont, P.A., Winston-Salem, North Carolina
  - Central Ohio Endoscopy Center LLC, Columbus, Ohio
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Integris Baptist Office, Oklahoma City, Oklahoma
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Essential Medical Research, Tulsa, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Gastroenterology Associates P.A., Greenville, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - West Texas Clinical Research, Lubbock, Texas
  - Victoria Gastroenterology, Richmond, Texas
  - Gastroenterology Clinic Of San Antonio P A, San Antonio, Texas
  - Wellness Clinical Research, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Care Access Research- Salt Lake City, Salt Lake City, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
- Australia (2):
  - Monash Health, Monash Medical Centre, Clayton
  - Coral Sea Clinical Research Institute, North Mackay
- Belgium (5):
  - OLV Ziekenhuis Aalst, Aalst
  - CHU Saint-Pierre, Brussels
  - Hopital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Algemeen Ziekenhuis Delta, Roeselare
- Bosnia and Herzegovina (6):
  - University hospital Clinical centre Banja Luka, Banja Luka
  - Clinical Center University of Sarajevo, Sarajevo
  - Polyclinic Dr. Al-Tawil, Sarajevo
  - General Hospital Tesanj, Tešanj
  - Plava poliklinika Tuzla, Tuzla
  - Cantonal Hospital Zenica, Zenica
- Brazil (28):
  - Universidade Estadual Paulista 'Julio De Mesquita Filho', Botucatu
  - CCB Centro Cardiologico de Brasilia Ltda - CCB Cardiologia, Brasília
  - Chronos Clinica Medica Ltda, Brasília
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - CDC - Centro Digestivo de Curitiba, Curitiba
  - Universidade Federal Do Ceara, Fortaleza
  - Centro de Estudos Clínicos do Interior Paulista - CECIP, Jaú
  - Cliged, Macaé
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Associacao dos Funcionarios Publicos do Estado do Rio Grande do Sul - Hospital Ernesto Dornelles, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Hospital das Clinicas - Universidade Federal de Pernambuco, Recife
  - Universidade Federal da Bahia - Hospital Professor Edgard Santos, Salvador
  - SER - Servicos Especializados em Reumatologia da Bahia, Salvador
  - Pesquisare Saude, Santo André
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Kaiser Hospta, São José do Rio Preto
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - BR TRIALS Ensaios Clinicos e Consultoria Ltda, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Hepatogastro, São Paulo
  - Fundacao Universidade Federal do Piaui - Universidade Federal do Piaui, Teresina
  - Integral Centro de Pesquisas Clinicas, Votuporanga
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
- China (26):
  - The Affiliated Hospital of Bengbu Medical College, Bengbu
  - Xiangya Hospital Central South University, Changsha
  - The second Xiangya Hospital of Central South University, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - Chongqing Medical University, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Guangzhou Medical University, Guangzhou
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Nanjing 1st Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Hospital of Quanzhou, Quanzhou
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - The first affiliated hospital of suzhou University, Suzhou
  - Wuxi People s Hospital, Wuxi
  - Yangzhou First People's Hospital, Yangzhou
  - ZhuZhou Central Hospital, Zhuzhou
- Croatia (4):
  - Opca bolnica Bjelovar, Bjelovar
  - University Hospital Center Split, Split
  - Opca bolnica Zadar, Zadar
  - Poliklinika Solmed, Zagreb
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Oblastni nemocnice Kladno a.s., Kladno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Nemocnice Slany, Slaný
- Denmark (2):
  - Sydvestjysk Sygehus, Esbjerg
  - Nordsjaellands Hospital - Hillerod, Hilleroed
- France (11):
  - Centre Hospitalier de la Cote Basque, Bayonne
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Hopital Louis Mourier, Colombes
  - CHU de Nantes hotel Dieu, Nantes
  - CHU de Nice Hopital de l Archet, Nice
  - Hôpital Bichat, Paris
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - Hôpital Robert Debré, Reims
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHRU Strasbourg, Strasbourg
  - CHU Rangueil, Toulouse
- Germany (13):
  - Charite Universitatsmedizin Berlin, Campus Mitte (CCM) Allergie Center, Berlin
  - DRK Kliniken Westend, Berlin
  - Krankenhaus Waldfriede Mitte, Berlin
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Evangelisches Krankenhaus Kalk, Cologne
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - MVZ Sanaklinikum Duisburg, Duisburg
  - BSF Studiengesellschaft, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Praxisgemeinschaft Jerichow, Jerichow
  - Gastroenterologische Spezialpraxis - Berlin-Karlshorst, Karlshorst
  - Universitaetsklinikum Mannheim, Mannheim
  - Tumorzentrum Nordthüringen Medizinisches Versorgungszentrum, Nordhausen
- Hungary (10):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Egyesített Szent István és Szent László Kórház, Budapest
  - Eszak Kozep budai Centrum Uj Szent Janos Korhaz es Szakrendelo Budai Csaladkozpontu, Budapest
  - Mh Egészségügyi Központ, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Mohacsi Korhaz, Mohács
  - Pecsi Tudomanyegyetem Orvostudomanyi Es Egeszsegtudomanyi Centrum, I. Belgyogyaszati Klinika, Pécs
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Israel (5):
  - Haemek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh Medical Center, Tzrifin
- Italy (3):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Istituto Clinico Humanitas Rozzano, IRCCS, Milan
  - Università Campus Biomedico di Roma, Roma
- Japan (42):
  - Juntendo University Hospital, Bunkyō City
  - Ginza central clinic, Chūōku
  - Fukui Prefectural Hospital, Fukui-ken
  - Fukuoka University Hospital, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - National Hospital Organization Fukuyama Medical Center, Fukuyama
  - Gamagori City Hospital, Gamagōri
  - Gunma University Hospital, Gunma
  - Hachinohe City Hospital, Hachinohe
  - Hamamatsu University Hospital, Hamamatsu
  - Matsuda Hospital, Hamamatsu
  - National Hospital Organization Mito Medical Center, Higashi-Ibaraki
  - Kure Kyosai Hospital, Hiroshima
  - National Hospital Organization Shikoku Cancer Center, Iizuka-shi
  - Kagoshima University Hospital, Kagoshima
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Kyushu Rosai Hospital, Kitakyushu
  - Kobe University Hospital, Kobe
  - Yamanashi Prefectural Central Hospital, Kofu
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Hidaka Coloproctologic Clinic, Kurume
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Iwate Medical University Hospital, Morioka
  - Nagasaki University Hospital, Nagasaki
  - Yokoyama IBD Clinic, Nagoya
  - University of the Ryukyus Hospital, Nakagami-gun
  - Niigata University Medical And Dental Hospital, Niigata
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Kinshukai Infusion Clinic, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Japanese Red Cross Osaka Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Oita Red Cross Hospital, Ōita
  - Shiga University of Medical Science Hospital, Ōtsu
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Takagi Clinic, Sendai
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun
  - Tokyo Medical University Hospital, Tokyo
  - Toyota Kosei Hospital, Toyota
  - Yokohama City University Medical Center, Yokohama
- Jordan (6):
  - Khalidi Hospital and Medical Center, Amman
  - The Speciality Hospital (TSH) / Advanced Clinical Center, Amman
  - Istiklal Hospital, Amman
  - Abdali Hospital, Amman
  - Irbid Specialty Hospital, Irbid
  - King Abdullah University Hospital, Irbid
- Lithuania (2):
  - Lietuvos sveikatos mokslų universiteto ligoninė Kauno klinik, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Public Institution, Vilnius
- Malaysia (5):
  - Hospital Sultanah Aminah, Johor Bharu
  - Hospital University Sains Malaysia, Kota Bharu
  - Hospital Raja Permaisuri Bainun, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Poland (44):
  - Gastromed Kralisz Romatowski Stachurska Sp. j., Bialystok
  - 10 Wojskowy Szpital Kliniczny z Poliklinika, SP ZOZ, Bydgoszcz
  - Centrum Medyczne Lukamed, Chojnice
  - Sahlgrenska University Hospital, Chrzanów
  - Private Practice - Dr. Krzysztof Cymerman, Gdynia
  - Centrum Medyczne Clw-Med Aneta Cichomska i Joanna Luka-Wendrowska sp.j., Grudziądz
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne ProMiMed, Krakow
  - AmiCare Centrum Medyczne, Lodz
  - IP Clinic Sp. z o.o., Lodz
  - Centrum Medyczne Med Gastr, Lodz
  - ETG Lublin, Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej, Lublin
  - Allmedica, Nowy Targ
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Twoja Przychodnia, Opole
  - Centrum Medyczne, Piotrkow Trybunalski
  - EMC Instytut Medyczny SA PL CERTUS, Poznan
  - Synexus Polska Sp z o o, Poznan
  - Twoja Przychodnia, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Centrum Medyczne Promed, Skorzewo
  - Endoskopia Sp z o.o., Sopot
  - Kiepury Clinic, Sosnowiec
  - KO Med Centrum Medyczne, Straszów
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Sonomed Sp. z o.o., Szczecin
  - GASTROMED Kopon Zmudzinski i wspolnicy SP j Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - H-T Centrum Medyczne Endoterapia, Tychy
  - Centrum Zdrowia Matki Dziecka i Mlodziezy, Warsaw
  - Endoterapia, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - NZOZ Vivamed, Warsaw
  - Gabinety Lekarskie Bodyclinic, Warsaw
  - IBD Point Profesor Kierkus, Warsaw
  - Centrum Zdrowia Tuchow, Wierzchosławice
  - Melita Medical Sp. z o.o., Wroclaw
  - Centrum Medyczne Melita Medical, Wroclaw
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego, Wroclaw
  - Przychodnia Vistamed, Wroclaw
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o. Szpital Specjalistyczny Barska, Włocławek
  - ETG Zamosc, Zamość
- Slovakia (3):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - ENDOMED s.r.o, Košice
  - GASTRO I. s.r.o., Prešov
- South Korea (18):
  - Kyungpook National University Chilgok Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - DongA Medical Center, Busan
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea Seoul St.Mary's Hospital, Daejeon
  - Kyung Hee University Hospital, Dongdaemun-gu
  - Dongguk University Ilsan Hospital, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University College of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Christian Hospital, Wŏnju
  - Ewha Womans University Mokdong Hospital, Yangch’ŏn-gu
- Spain (6):
  - Hosp. de Cabuenes, Gijón
  - Hosp. Gral. Juan Ramon Jimenez, Huelva
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Virgen Macarena, Seville
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. de La Marina Baixa, Villajoyosa
- Taiwan (5):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaoshiung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Division of Infectious Diseases, Taipei
  - Taipei Medical University, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (8):
  - Ankara Numune Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe University Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Acibadem Fulya Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis University, Samsun
  - Bülent Ecevit Üniversitesi Sağlık Uygulama ve Araştırma Hastanesi, Zonguldak

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Hart A, Panaccione R, Steinwurz F, Danese S, Hisamatsu T, Cao Q, Ritter T, Seidler U, Olurinde M, Vetter ML, Yee J, Yang Z, Wang Y, Johanns J, Han C, Sahoo A, Terry NA, Sands BE, D'Haens G; GRAVITI Study Group. Efficacy and Safety of Guselkumab Subcutaneous Induction and Maintenance in Participants With Moderately to Severely Active Crohn's Disease: Results From the Phase 3 GRAVITI Study. Gastroenterology. 2025 Aug;169(2):308-325. doi: 10.1053/j.gastro.2025.02.033. Epub 2025 Mar 18. PMID 40113101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 350 participants randomized (1:1:1) to 1 of 3 treatments, 3 participants were excluded from all analysis sets due to non-compliance with Good Clinical Practice (GCP) guidance at 1 study site. Hence 347 participants were included in full analysis set. Study included a 24 week (wk) main treatment (12-wk induction followed by 12-wk maintenance) period followed by extension treatment period. In extension period, participants continued same maintenance dose regimen they received at Week 24.
Pre-assignment Details: Results through the Week 48 visit (cutoff date of 01 March 2024) are reported. Results of remaining duration of the study will be reported after study completion.
Groups:
- Placebo: Participants received placebo matched to guselkumab 400 milligrams (mg) subcutaneous (SC) injection at Weeks 0, 4, and 8 followed by placebo matched to guselkumab 200 mg SC injection every 4 weeks from Week 12 through Week 48 and placebo matched to guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48. Participants who met at least one of the rescue criteria (Crohn's Disease Activity Index [CDAI] score greater than [>] 220 and less than [<] 70-point reduction from baseline CDAI score at both Weeks 12 and 16 or at least 50 percent [%] increase in Simple Endoscopic Score for Crohn's Disease [SES-CD] from baseline at Week 12) at Week 16 received rescue treatment: guselkumab 400 mg SC injection at Weeks 16, 20, and 24 along with placebo matched to guselkumab 100 mg SC injection on Weeks 16 and 24 followed by guselkumab 100 mg SC injection every 8 weeks from Week 32 through Week 48 and placebo matched to guselkumab 200 mg SC injection every 4 weeks from Week 28 through Week 48.
- Guselkumab 400 mg + 100 mg: Participants received guselkumab 400 mg SC injection at Weeks 0, 4, and 8, followed by guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48 and a placebo matched to guselkumab 200 mg SC injection every 4 weeks from Week 12 through Week 48. Participants who met at least one of the rescue criteria (CDAI score >220 and <70-point reduction from baseline CDAI score at both Weeks 12 and 16 or at least 50% increase in SES-CD from baseline at Week 12) at Week 16 received rescue treatment (sham): continued receiving guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48, along with placebo matched to guselkumab 400 mg SC injection on Weeks 16, 20 and 24, and placebo matched to guselkumab 200 mg SC injection every 4 weeks from Week 28 through Week 48.
- Guselkumab 400 mg + 200 mg: Participants received guselkumab 400 mg SC injection at Weeks 0, 4, and 8, followed by guselkumab 200 mg SC injection every 4 weeks from Week 12 through Week 48, and a placebo matched to guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48. Participants who met at least one of the rescue criteria (CDAI score >220 and <70-point reduction from baseline CDAI score at both Weeks 12 and 16 or at least 50% increase in SES-CD from baseline at Week 12) at Week 16 received rescue treatment: (sham): continued receiving guselkumab 200 mg SC injection every 4 weeks from Week 16 through Week 48, along with placebo matched to guselkumab 200 mg SC injection on Weeks 16, 20 and 24 and placebo matched to guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48.
Period: Overall Study
Arm/Group | Placebo | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg
Started | 118 | 117 | 115
Treated | 117 | 115 | 115
Participants Who Met at Least 1 Rescue Criteria at Week 16 | 44 | 14 | 14
Completed ('Completed' signified all participants who completed study through Week 48 at cutoff date (01-Mar-2024).) | 99 | 110 | 114
Not Completed | 19 | 7 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Withdrawal by Subject | 15 | 3 | 1
Not completed — GCP non-compliance | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were presented for full analysis set (FAS) which included all randomized participants who received at least 1 dose of study intervention.
Groups:
- Placebo: Participants received placebo matched to guselkumab 400 milligrams (mg) subcutaneous (SC) injection at Weeks 0, 4, and 8 followed by placebo matched to guselkumab 200 mg SC injection every 4 weeks from Week 12 through Week 48 and placebo matched to guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48. Participants who met at least one of the rescue criteria (CDAI score >220 and <70-point reduction from baseline CDAI score at both Weeks 12 and 16 or at least 50% increase in SES-CD from baseline at Week 12) at Week 16 received rescue treatment: guselkumab 400 mg SC injection at Weeks 16, 20, and 24 along with placebo matched to guselkumab 100 mg on Week 16 and 24 followed by guselkumab 100 mg SC injection every 8 weeks from Week 32 through Week 48 and placebo matched to guselkumab 200 mg every 4 weeks from Week 28 through Week 48.
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg | Total
Number analyzed (Participants) | 117 | 115 | 115 | 347
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 114 | 113 | 111 | 338
  >=65 years | 3 | 2 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 45 | 144
  Male | 67 | 66 | 70 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 8 | 27
  Not Hispanic or Latino | 93 | 94 | 98 | 285
  Unknown or Not Reported | 15 | 11 | 9 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 28 | 26 | 22 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 4 | 9
  White | 71 | 79 | 79 | 229
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 10 | 10 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 1 | 0 | 1 | 2
  Bosnia | 3 | 4 | 4 | 11
  BRAZIL | 13 | 12 | 7 | 32
  CHINA | 19 | 16 | 16 | 51
  CROATIA | 0 | 1 | 2 | 3
  CZECH REPUBLIC | 5 | 7 | 2 | 14
  FRANCE | 5 | 3 | 3 | 11
  GERMANY | 4 | 8 | 1 | 13
  HUNGARY | 4 | 3 | 3 | 10
  ISRAEL | 0 | 0 | 1 | 1
  ITALY | 0 | 1 | 1 | 2
  JAPAN | 5 | 1 | 0 | 6
  JORDAN | 15 | 8 | 9 | 32
  LITHUANIA | 1 | 0 | 2 | 3
  MALAYSIA | 0 | 1 | 2 | 3
  NEW ZEALAND | 0 | 1 | 1 | 2
  POLAND | 27 | 28 | 33 | 88
  SLOVAKIA | 1 | 4 | 4 | 9
  SOUTH KOREA | 2 | 6 | 3 | 11
  SPAIN | 1 | 3 | 1 | 5
  TAIWAN | 2 | 0 | 1 | 3
  TURKEY | 1 | 3 | 1 | 5
  UNITED STATES | 8 | 5 | 17 | 30
AgeContinuous [Mean (Standard Deviation); unit: years] | 36 (12.71) | 37.4 (13.32) | 39.1 (12.56) | 37.5 (12.89)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 12
Description: Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) and a decrease in total CDAI score over time indicates improvement in disease activity.
Time Frame: At Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study intervention. As prespecified in Statistical Analysis Plan (SAP), for this outcome measure (OM), combined data for both guselkumab treatment groups were collected and analyzed because they received the same regimen of guselkumab 400 mg SC at Weeks 0, 4, and 8.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Participants received placebo matched to guselkumab 400 milligrams (mg) subcutaneous (SC) injection at Weeks 0, 4, and 8 followed by placebo matched to guselkumab 200 mg SC injection every 4 weeks from Week 12 through Week 48 and placebo matched to guselkumab 100 mg SC injection every 8 weeks from Week 16 through Week 48. Participants who met at least one of the rescue criteria (Crohn's Disease Activity Index [CDAI] score greater than [>] 220 and less than [<] 70-point reduction from baseline CDAI score at both Weeks 12 and 16 or at least 50 percent [%] increase in Simple Endoscopic Score for Crohn's Disease [SES-CD] from baseline at Week 12) at Week 16 received rescue treatment: guselkumab 400 mg SC injection at Weeks 16, 20, and 24 along with placebo matched to guselkumab 100 mg on Week 16 and 24 followed by guselkumab 100 mg SC injection every 8 weeks from Week 32 through Week 48 and placebo matched to guselkumab 200 mg every 4 weeks from Week 28 through Week 48.
- Combined: Guselkumab 400 mg: Participants of arm "Guselkumab 400 mg + 100 mg" and "Guselkumab 400 mg + 200 mg" received guselkumab 400 mg SC injections at Week 0, 4, and 8.
Arm/Group | Placebo | Combined: Guselkumab 400 mg
Number analyzed (Participants) | 117 | 230
Percentage of participants | 21.4 [13.9 to 28.8] | 56.1 [49.7 to 62.5]
Statistical Analysis 1: Comparison: Placebo vs Combined: Guselkumab 400 mg; Test type: Superiority; p < 0.001, Mantel Haenszel; Mantel-Haenszel stratum weights and the Sato variance estimator; Adjusted treatment difference:percentage = 34.9, 95% CI 2-sided [25.1 to 44.6]

2. Primary Outcome: Percentage of Participants Who Achieved Endoscopic Response at Week 12
Description: Percentage of participants who achieved endoscopic response at Week 12 were reported. Endoscopic response was defined as greater than or equal to (>=) 50 percent (%) improvement from baseline in the Simple Endoscopic Score for Crohn's Disease (SES-CD) score. SES-CD evaluated 4 endoscopic components (presence and size of ulcer, extent of ulcerated surface, extent of affected surface, and presence and type of narrowing) across 5 ileocolonic segments (ileum, right colon, transverse colon, left colon, and rectum), each scored from 0 (best) to 3 (worst) for each segment except narrowing component for which the maximum total score (that is, stricturing) was 11 points. The total SES-CD score was the sum of all the component scores across all the segments and it ranged from 0 (best) to 56 (worst), where higher scores indicated more severe disease.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined: Guselkumab 400 mg
Number analyzed (Participants) | 117 | 230
Percentage of participants | 21.4 [13.9 to 28.8] | 41.3 [34.9 to 47.7]
Statistical Analysis 1: Comparison: Placebo vs Combined: Guselkumab 400 mg; Test type: Superiority; p < 0.001, Mantel Haenszel; Mantel-Haenszel stratum weights and the Sato variance estimator; Adjusted treatment difference:percentage = 19.9, 95% CI 2-sided [10.2 to 29.6]

3. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 24
Description: Percentage of participants who achieved clinical remission at Week 24 were reported. Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) and a decrease in total CDAI score over time indicates improvement in disease activity.
Time Frame: At Week 24
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg
Number analyzed (Participants) | 117 | 115 | 115
Percentage of participants | 21.4 [13.9 to 28.8] | 60.9 [51.9 to 69.8] | 58.3 [49.2 to 67.3]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 400 mg + 200 mg; Test type: Superiority; p < 0.001, Mantel Haenszel; Mantel-Haenszel stratum weights and the Sato variance estimator; Adjusted treatment difference:percentage = 37.0, 95% CI 2-sided [25.6 to 48.4]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 400 mg + 100 mg; Test type: Superiority; p < 0.001, Mantel Haenszel; Mantel-Haenszel stratum weights and the Sato variance estimator; Adjusted treatment difference:percentage = 39.3, 95% CI 2-sided [28.0 to 50.7]

4. Secondary Outcome: Percentage of Participants Who Achieved Patient-reported Outcome (PRO)-2 Remission at Week 12
Description: Percentage of participants who achieved PRO-2 remission at Week 12 were reported. PRO-2 remission was defined as an abdominal pain (AP) mean daily score <=1, and stool frequency (SF) mean daily score <=3, and no worsening of AP or SF from baseline. Mean daily AP score based on the CDAI was defined as the sum of abdominal pain/cramps ratings in the previous 7 days in a diary card divided by the total number of days assessments were performed. Average daily SF score based on the CDAI was defined as the sum of number of liquid or very soft stools in the previous 7 days in a diary card divided by the total number of days assessments were performed. Mean daily SF and AP scores at a scheduled visit were not calculated if total number of days of assessment was less than 5. Higher PRO-2 scores indicated more severe disease.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined: Guselkumab 400 mg
Number analyzed (Participants) | 117 | 230
Percentage of participants | 17.1 [10.3 to 23.9] | 49.1 [42.7 to 55.6]
Statistical Analysis 1: Comparison: Placebo vs Combined: Guselkumab 400 mg; Test type: Superiority; p < 0.001, Mantel Haenszel; Mantel-Haenszel stratum weights and the Sato variance estimator; Adjusted treatment difference:percentage = 32.1, 95% CI 2-sided [22.9 to 41.2]

5. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response at Week 12
Description: Clinical response was defined as a decrease from baseline in CDAI score >= 100 points or CDAI score < 150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) and a decrease in total CDAI score over time indicates improvement in disease activity.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined: Guselkumab 400 mg
Number analyzed (Participants) | 117 | 230
Percentage of participants | 33.3 [24.8 to 41.9] | 73.5 [67.8 to 79.2]
Statistical Analysis 1: Comparison: Placebo vs Combined: Guselkumab 400 mg; Test type: Superiority; p < 0.001, Mantel Haenszel; Mantel-Haenszel stratum weights and the Sato variance estimator; Adjusted treatment difference:percentage = 40.3, 95% CI 2-sided [29.9 to 50.7]

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Through Week 48
Description: Percentage of participants with TEAEs through Week 48 were reported. An adverse event (AE) was any untoward medical occurrence in a clinical study participant participating in a clinical study and does not necessarily have a causal relationship with the study drug. An AE that occurred at or after the initial administration of study drug (Week 0) through data cutoff of Week 48 was considered treatment-emergent.
Time Frame: Placebo, Guselkumab 400 mg + 100 mg, and Guselkumab 400 mg + 200 mg: From Week 0 up to Week 48; Placebo arm subset - Rescue Treatment: From Week 16 up to Week 48
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab: Participants randomized to placebo arm who met at least one of the rescue criteria (CDAI score >220 and <70-point reduction from baseline CDAI score at both Weeks 12 and 16 or at least 50% increase in SES-CD from baseline at Week 12) at Week 16 received rescue treatment: guselkumab 400 mg SC injection at Weeks 16, 20, and 24 along with placebo matched to guselkumab 100 mg on Week 16 and 24 followed by guselkumab 100 mg SC injection every 8 weeks from Week 32 through Week 48 and placebo matched to guselkumab 200 mg every 4 weeks from Week 28 through Week 48. For this arm, data were collected and analyzed after the participants of arm "Placebo" crossed over to receive rescue treatment with guselkumab.
Arm/Group | Placebo | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg | Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab
Number analyzed (Participants) | 117 | 115 | 115 | 44
Percentage of participants | 65.8 | 82.6 | 80.0 | 75.0

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) Through Week 48
Description: Percentage of participants with TESAEs through Week 48 were reported. An SAE was any untoward medical occurrence in a clinical study participant resulting in any of the following outcomes or was deemed significant for any other reason: death, life-threatening (immediate risk of dying), initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect. An AE does not necessarily have a causal relationship with the study drug. Any SAE that occurred at or after the initial administration of study drug (Week 0) through the data cutoff of Week 48 was considered treatment-emergent.
Time Frame: as for outcome 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg | Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab
Number analyzed (Participants) | 117 | 115 | 115 | 44
Percentage of participants | 13.7 | 13.0 | 7.8 | 2.3

8. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug Through Week 48
Description: Percentage of participants with TEAEs leading to discontinuation of study drug through Week 48 were reported. An adverse event (AE) was any untoward medical occurrence in a clinical study participant participating in a clinical study and does not necessarily have a causal relationship with the study drug. An AE that occurred at or after the initial administration of study drug (Week 0) through data cutoff of Week 48 was considered treatment-emergent.
Time Frame: as for outcome 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg | Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab
Number analyzed (Participants) | 117 | 115 | 115 | 44
Percentage of participants | 8.5 | 3.5 | 2.6 | 2.3

ADVERSE EVENTS:
Time Frame: For arms Placebo, Guselkumab 400 mg + 100 mg, and Guselkumab 400 mg + 200 mg: From Week 0 up to Week 48; Placebo arm subset - Rescue Treatment: From Week 16 up to Week 48
Description: Safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Placebo | Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab | Guselkumab 400 mg + 100 mg | Guselkumab 400 mg + 200 mg
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/44 | 1/115 | 0/115
Serious Adverse Events (participants affected / at risk) | 16/117 | 1/44 | 15/115 | 9/115
Other Adverse Events (participants affected / at risk) | 57/117 | 19/44 | 65/115 | 68/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab (N=44) | Guselkumab 400 mg + 100 mg (N=115) | Guselkumab 400 mg + 200 mg (N=115)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Thyroid Cyst (Endocrine disorders) | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 7 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gastrointestinal Anastomotic Stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intraductal Papilloma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Breast Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Placebo Arm Subset (Rescue Treatment): Placebo to Guselkumab (N=44) | Guselkumab 400 mg + 100 mg (N=115) | Guselkumab 400 mg + 200 mg (N=115)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 8 | 2
Abdominal Pain (Gastrointestinal disorders) | 7 | 3 | 10 | 14
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 4 | 1
Crohn's Disease (Gastrointestinal disorders) | 17 | 3 | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 6 | 4
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 5
Fatigue (General disorders) | 0 | 0 | 3 | 4
Pyrexia (General disorders) | 8 | 2 | 3 | 6
Covid-19 (Infections and infestations) | 8 | 1 | 11 | 11
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 4
Gastroenteritis (Infections and infestations) | 1 | 2 | 4 | 1
Influenza (Infections and infestations) | 5 | 1 | 6 | 6
Nasopharyngitis (Infections and infestations) | 6 | 3 | 8 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 5 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 8 | 15 | 15
Aspartate Aminotransferase Increased (Investigations) | 4 | 1 | 2 | 2
White Blood Cell Count Decreased (Investigations) | 1 | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 6 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 5 | 1 | 7 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT05197049/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT05197049/SAP_001.pdf